CLINICAL TRIAL: NCT04563806
Title: A Pilot Study to Evaluate the Safety of MRI Compatible Hardware for Intraoperative MRI-Based Image Guidance for Spinal Procedures
Brief Title: Safety of MRI Compatible Hardware for MRI-based Image Guidance During Spine Surgery
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Per PI
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-0663; NCI-2020-03700 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0663 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-10; First posted 2020-09-24 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Thoracic Spine Neoplasm
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device feasibility (MRI-guided surgery) (Experimental): Patients undergo standard of care spine surgery with MRI-based image guidance.
  Interventions: Device: Magnetic Resonance Imaging; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Undergo MRI-guided surgery
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Therapeutic Conventional Surgery — Undergo spinal surgery

SUMMARY:
This trial investigates the safety and accuracy of using 2 pieces of hardware (a clamp and a needle) that are able to be used with magnetic resonance imaging (MRI) during spinal surgery. During a standard spinal surgery, a computed tomography (CT) scan is used to help plan the placement of surgical instruments used during the procedure or for needle biopsies. Then, the patient is moved to the MRI. For this study, the patient is able to stay in place as the hardware used in this study is able to work with the MRI. Using MRI compatible hardware may allow for an extra degree of safety and facilitate better surgical workflow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To document the safety of utilizing MRI compatible hardware for intraoperative MRI-based image guidance to perform percutaneous spinal procedures.

SECONDARY OBJECTIVE:

I. To determine the accuracy of the MRI-based image guidance.

OUTLINE:

Patients undergo standard of care spine surgery with MRI-based image guidance.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing percutaneous spinal procedures requiring image guidance at MD Anderson
* Age > 18 years old. (The indication for this technique is controversial in skeletally immature patients.)
* All diagnoses are eligible
* Vertebral body site to be treated located from T2 to T12
* Signed informed consent

Exclusion Criteria:

* Requires open spinal procedure or a percutaneous procedure without the use of image guidance
* Unable to tolerate general anesthesia and prone position
* Unable to undergo MRI scan of the spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative adverse events | During surgery
  Safety will be assessed as a dichotomous variable. Frequencies and descriptive statistics of the outcomes under study will be performed. 95% confidence intervals will be computed. Other ad-hoc analyses may be performed as well.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio E Tatsui, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org